CLINICAL TRIAL: NCT04549298
Title: Assessment of the Possible Association Between Left Ventricular Diastolic Dysfunction and Carotid Atherosclerosis and Brain White Matter Damage
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Principal Investigator, Giuseppe Lembo, Full Professor, MD, PhD, Neuromed IRCCS
Other Study IDs: LMB09
Record Dates: First submitted 2020-09-08; First posted 2020-09-16 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Left Ventricular Diastolic Dysfunction
Keywords: Diastolic dysfunction; White matter hyperintensities; Carotid atherosclerosis
MeSH Terms: conditions — Ventricular Dysfunction, Left; Carotid Artery Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with grade 2 and 3 LV diastolic dysfunction: Patients with high filling pressure
  Interventions: Other: No interventions
- Patients with normal and grade 1 LV diastolic dysfunction: Patients with normal filling pressure
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions — No interventions - observational study

SUMMARY:
Left ventricular diastolic dysfunction is caused by impaired relaxation and increased left ventricular stiffness with a consequent increase in filling pressures. Currently, it is possible to classify it in 3 grades: grade 1 with normal filling pressures, grade 2 and grade 3 with high pressures. Diastolic dysfunction is closely associated with several risk factors such as hypertension, diabetes, and obesity, as well as the risk of heart failure, cardiovascular events, and death. In the field of cerebrovascular diseases, however, diastolic dysfunction is still being researched. Thus, this study aims to: 1) evaluate the white matter hyperintensities volume in association with the increase of diastolic dysfunction and filling pressures 2) evaluate the possible association with carotid atherosclerosis in case of brain damage caused by dysfunction diastolic 3) understand the mechanism of damage caused by left ventricular diastolic dysfunction on the cerebrovascular system. In order to do this, this study proposes to evaluate in a cohort of patients, between 35 and 65 years, the possible association of diastolic dysfunction with lesions on the cerebrovascular system in a future view of new marker of brain damage and new modifiable risk factor.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 35 and ≤ 65 years
* written informed consent

Exclusion Criteria:

* previous stroke or TIA
* arrhythmia or severe cardiac disease
* renal disease
* psychiatric disease
* neurological or neurodegenerative disease
* dementia
* previous carotid artery stenting or carotid surgery
* inability to be subjected MRI analysis

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be selected from patients attending the Department of AngioCardioNeurology of the IRCCS Neuromed, accordingly to the following inclusion/exclusion criteria. Approximately 88 subjects of both genders will be included in the study.
Sampling Method: Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Measurement of white matter hyperintensities volume | At Enrollment
  Brain MRI

SECONDARY OUTCOMES:
Detection of plaques and carotid atherosclerosis | At Enrollment
  Ultrasound of the supraortic trunks
Characterization of cardiac overload with blood markers | At Enrollment
  NT-proBNP
Detection of cognitive decline by decrease of MoCA score | At Enrollment
  Cognitive tests

IPD SHARING:
Plan to Share IPD: No